CLINICAL TRIAL: NCT00021541
Title: A Phase II Randomized, Cross-Over, Double-Blinded, Placebo-Controlled Trial of the Farnesyltransferase Inhibitor R115777 in Pediatric Patients With Neurofibromatosis Type I and Progressive Plexiform Neurofibromas
Brief Title: R115777 to Treat Children With Neurofibromatosis Type 1 and Progressive Plexiform Neurofibromas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Brigitte Widemann, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 010222; 01-C-0222; NCT00029354 (obsolete NCT alias)
Record Dates: First submitted 2006-06-19; First posted 2001-07-23 (Estimated); Results first posted 2012-09-17 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-03

CONDITIONS: Neurofibroma, Plexiform; Neurofibromatosis Type I
Keywords: Surrogate Markers; 3-Dimensional Magnetic Resonance Imaging (MRI); Natural History of Neurofibromatosis Type 1 (NF1); Tumor Tissue Bank; Neurofibromatosis; NF1; Neurofibromatosis Type 1; Plexiform Neurofibroma; Neurofibroma
MeSH Terms: conditions — Neurofibroma, Plexiform; Neurofibromatosis 1; Neurofibromatoses; Neurofibroma | interventions — tipifarnib

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tipifarnib (R11577)-Arm I (Experimental): Patients receive oral R115777 (Tipifarnib) first followed by placebo. 200 mg/m^2/dose BSA every 12 hours by mouth (po)on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: tipifarnib
- Placebo-Arm II (Placebo Comparator): Patients receive oral placebo first followed by R115777 (Tipifarnib). 200 mg/m^2/dose BSA every 12 hours by mouth (po)every 12 hours on days 1-21. Courses repeat as in arm I.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: tipifarnib — Given orally, 200 mg/m^2/dose BSA every 12 hours by mouth (po) daily x 21 days, Course is every 28 days
  Other Names: R115777
  Arms: Tipifarnib (R11577)-Arm I
Other: placebo — Patients receive oral placebo every 12 hours on days 1-21. Courses repeat as in arm I.
  Arms: Placebo-Arm II

SUMMARY:
This study will examine whether the experimental drug R115777 (Tipifarnib) can shrink or slow the growth of plexiform neurofibromas in children and young adults with neurofibromatosis type 1 (NF1) and determine what side effects are related to treatment. Plexiform tumors arise from nerves; the only effective treatment is surgical removal. Often, however, not all the tumors can be removed, because of their number or location.

Patients with NF1 have a reduced amount of the protein neurofibromin. Neurofibromin is thought to help control the activity of another protein, called ras, which regulates cell growth. Too little neurofibromin, therefore, may allow for uncontrolled cell growth and tumor formation. R115777 interferes with the function of the ras and other proteins. In test tube and animal studies, R115777 has blocked the growth of cancer cells. This study will examine whether the drug is effective against plexiform tumors.

Patients with NF1 and progressive plexiform neurofibromas between 3 and 25 years of age may be eligible for this study. Patients whose tumors can be successfully removed surgically may not participate in this study. Candidates are screened with a medical history and physical and eye examinations, blood and urine tests, and magnetic resonance imaging (MRI). Photographs are taken of tumors visible on the body surface.

Study participants are randomly assigned to receive either R115777 or placebo (an inactive substance). They take R115777 or placebo tablets every 12 hours for 21 days, followed by a 7-day rest period. This constitutes one 28-day treatment cycle. Treatment continues for as long as the tumors remain stable or shrink and side effects are tolerable. The treatment is switched (for example, from placebo to R115777) or stopped if the tumors grow or if side effects become unacceptable. Patients (or their parents) keep a record of side effects.

For the first 3 treatment cycles, patients have a physical examination and blood tests every other week. Blood tests are also done before starting treatment, and at one time point after at least 14 days of treatment to measure the effect of R115777 on proteins in blood cells. A blood sample is obtained before starting treatment and before cycles 4, 7 and 10 and then after every 6 cycles to measure the level of a substance called nerve growth factor. The analysis of nerve growth factor is used to determine if it can predict which patients might be at risk of developing side effects from R115777.

DETAILED DESCRIPTION:
R115777 (Tipifarnib) is a farnesyltransferase inhibitor that blocks the post-translational isoprenylation of ras and other farnesylated proteins. The ras proteins are integral in cell signaling pathways, and farnesylation is essential for the function of both mutant and non-mutant ras proteins. Patients with neurofibromatosis type 1 (NF1) have an increased risk of developing tumors of the central and peripheral nervous system, and there are no standard treatment options, other than surgery, available for these tumors. Neurofibromin, which is the product of the NF1 gene, contains a domain with significant homology to ras GTPase-activating proteins (GAP). Although NF1 patients lack germline ras mutations, the decreased levels of neurofibromin have been shown to be associated with a constitutively activated ras-GTP status. Thus, upstream inhibition of ras farnesylation may inhibit growth of tumors in NF1 patients. A randomized, cross-over, double-blinded, placebo-controlled pediatric phase II trial of oral R115777 will be performed in children and young adults with NF1, who have progressive, plexiform neurofibroma(s) to determine the effect of this novel anticancer drug on the rate of growth of neurofibromas. The endpoint of the trial is time to progression. R115777 will be administered orally at a dose of 200 mg/m(2) twice daily for cycles of 21 days followed by a 7 day rest period based on the results of our prior pediatric phase I trial.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age: 3 years and 25 years of age.

Diagnosis: Patients with neurofibromatosis type 1 (NF1) and progressive plexiform neurofibromas that have the potential to cause significant morbidity, such as (but not limited to) head and neck lesions that could compromise the airway or great vessels, brachial or lumbar plexus lesions that could cause nerve compression and loss of function, lesions that could result in major deformity (e.g., orbital lesions), lesions of the extremity that cause limb hypertrophy or loss of function, and painful lesions.

Histologic confirmation of tumor is not necessary in the presence of consistent clinical and radiographic findings, clinically suspected.

In addition to plexiform neurofibroma(s), all study subjects must have at least one other diagnostic criteria for NF1 listed below (National Institutes of Health (NIH) Consensus Conference[9]):

1. Six or more cafe-au-lait spots (0.5 cm in prepubertal subjects or 1.5 cm in postpubertal subjects).
2. Freckling in the axilla or groin;
3. Optic glioma;
4. Two or more Lisch nodules;
5. A distinctive bony lesion (dysplasia of the sphenoid bone or dysplasia or thinning of long bone cortex);
6. A first degree relative with NF1.

In this study a plexiform neurofibroma is defined as a neurofibroma that has grown along the length of a nerve and may involve multiple fascicles and branches.

A spinal plexiform neurofibroma involves two or more levels with connection between the levels or extending laterally along the nerve.

Measurable disease: Patients must have measurable plexiform neurofibroma(s). For the purpose of this study a measurable lesion will be defined as a lesion of at least 3 cm measured in one dimension.

There must be evidence of recurrent or progressive disease as documented by an increase in size or the presence of new plexiform neurofibromas on MRI. Progression at the time of study entry is defined as:

1. A measurable increase of the plexiform neurofibroma (20% increase in the volume, or a 13% increase in the product of the two longest perpendicular diameters, or a 6% increase in the longest diameter) over the last two consecutive scans (magnetic resonance imaging (MRI) or computed tomography (CT)), or over the time period of approximately one year prior to evaluation for this study.
2. Patients who underwent surgery for a progressive plexiform neurofibroma will be eligible to enter the study after the surgery, provided the plexiform neurofibroma was incompletely resected and is measurable.

   Prior therapy: Patients with NF1 are eligible at the time of recurrence or progression of inoperable plexiform neurofibroma.

   A surgical consultation should be obtained prior to enrollment on the study to evaluate if tumor resection is a feasible option.

   Patients will only be eligible if complete tumor resection is not feasible, or if a patient with surgical option refuses surgery.

   Since there is no standard effective chemotherapy for patients with NF1 and progressive plexiform neurofibromas, patients may be treated on this trial without having received prior therapy.

   Patients must have recovered from the toxic effects of all prior therapy before entering this study.

   The Cancer Therapy Evaluation Program Common Toxicity Criteria (CTC) Version 2.0 will be used for toxicity assessment.

   A copy of the CTC version 2.0 can be downloaded from the CTEP home page: http://ctep.cancer.gov. Recovery is defined as a toxicity grade less than 2, unless otherwise specified in the Inclusion and Exclusion Criteria.

   Patients must have had their last dose of radiation therapy at least six weeks prior to study entry, and their last dose of chemotherapy at least four weeks prior to study entry.

   Patients who received growth colony stimulating factor (G-CSF) after the prior cycle of chemotherapy must be off G-CSF for at least one week prior to entering this study.

   Performance Status: Patients should have a life expectancy of at least 12 months and an Eastern Cooperative Oncology Group (ECOG) performance score of 0, 1, or 2.

   Patients who are wheelchair bound because of paralysis should be considered 'ambulatory' when they are up in their wheelchair.

   Hematologic Function: Patients must have an absolute granulocyte count 1,500/ uL, 9.0 gm/dl, and a platelet count 150,000/uL at study entry, and a normal fibrinogen.

   Hepatic Function: Patients must have a bilirubin within normal limits and serum glutamic pyruvic transaminase (SGPT) 2x upper limit of normal.

   Patients with Gilbert syndrome are excluded from the requirement of a normal bilirubin. (Gilbert syndrome is found in 3-10% of the general population, and is characterized by mild, chronic unconjugated hyperbilirubinemia in the absence of liver disease or overt hemolysis).

   Renal Function: Patients must have an age-adjusted normal serum creatinine OR a creatinine clearance (70 mL / min / 1.73 m^2).

   Informed Consent: All patients or their legal guardians (if the patient is less than 18 years old) must sign an institutional review board (IRB) approved document of informed consent (screening protocol) prior to performing studies obtained exclusively to determine patient eligibility.

   After confirmation of patient eligibility all patients or their legal guardians must sign the protocol specific informed consent to document their understanding of the investigational nature and the risk of this study before any protocol related studies are performed (other than the studies which were performed to determine patient eligibility).

   When appropriate pediatric patients will be included in all discussion. Per institutional guidelines, age appropriate assent forms for children from 7 through 12 years, and for children may be developed and, when appropriate, will be signed by the pediatric patients in order to obtain written assent.

   Durable Power of Attorney (DPA):

   All patients 18 years of age will be offered the opportunity to assign DPA so that another person can make decisions about their medical care if they become incapacitated or cognitively impaired.

   Ability to undergo MRI examinations.

   EXCLUSION CRITERIA:

   Pregnant or breast feeding females are excluded, because the toxic effects and pharmacology of R115777 in the fetus and newborn are unknown.

   Clinically significant unrelated systemic illness (serious infections or significant cardiac, pulmonary, hepatic or other organ dysfunction) which in the judgement of the Principal or Associate Investigator would compromise the patient's ability to tolerate R115777 or are likely to interfere with the study procedures or results.

   Prior treatment with greater than 1 prior myelosuppressive chemotherapy regimen.

   An investigational agent within the past 30 days.

   Evidence of an optic glioma, malignant glioma, malignant peripheral nerve sheath tumor or other cancer requiring treatment with chemotherapy or radiation therapy.

   Ongoing radiation therapy, chemotherapy, hormonal therapy directed at the tumor, or immunotherapy.

   Inability to return for follow-up visits or obtain follow-up studies required to assess toxicity and response to therapy.

   Prior treatment with R115777.

Ages: 3 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 62 (Actual)
Dates: Start 2001-07-17 (Actual); Primary Completion 2009-02-19 (Actual); Study Completion 2009-02-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Widemann, M.D., Principal Investigator — National Insitutes of Health, National Cancer Institute
Locations (12):
- United States (11):
  - University of Alabama at Birmingham (M1149), Birmingham, Alabama
  - Children's Hospital Los Angeles, CA (M1118), Los Angeles, California
  - Children's Memorial Hospital, Chicago, IL (M1484), Chicago, Illinois
  - Johns Hopkins Oncology Center (M1011), Baltimore, Maryland
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - The Children's Hospital, Dana-Farber Cancer Institute, Boston, MA (M1034), Boston, Massachusetts
  - St. Louis Children's Hospital, St. Louis, MO (M1123), St Louis, Missouri
  - SUNY Upstate Medical University, NY (M1303), Syracuse, New York
  - Cincinnati Children's Hospital (FWA 00002988), Cincinnati, Ohio
  - Childrens Hospital of Philadelphia, PA (M1257), Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, TX (M1060), Houston, Texas
- Klinikum Nord, Hamburg, Germany (FWA 00003228), Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bernards A. Neurofibromatosis type 1 and Ras-mediated signaling: filling in the GAPs. Biochim Biophys Acta. 1995 Jul 28;1242(1):43-59. doi: 10.1016/0304-419x(95)00003-x. No abstract available. PMID 7626654
- [Background] De Santis S, Pace A, Bove L, Cognetti F, Properzi F, Fiore M, Triaca V, Savarese A, Simone MD, Jandolo B, Manzione L, Aloe L. Patients treated with antitumor drugs displaying neurological deficits are characterized by a low circulating level of nerve growth factor. Clin Cancer Res. 2000 Jan;6(1):90-5. PMID 10656436
- [Background] Goldberg Y, Dibbern K, Klein J, Riccardi VM, Graham JM Jr. Neurofibromatosis type 1--an update and review for the primary pediatrician. Clin Pediatr (Phila). 1996 Nov;35(11):545-61. doi: 10.1177/000992289603501101. PMID 8953130
- [Result] Widemann BC, Dombi E, Gillespie A, Wolters PL, Belasco J, Goldman S, Korf BR, Solomon J, Martin S, Salzer W, Fox E, Patronas N, Kieran MW, Perentesis JP, Reddy A, Wright JJ, Kim A, Steinberg SM, Balis FM. Phase 2 randomized, flexible crossover, double-blinded, placebo-controlled trial of the farnesyltransferase inhibitor tipifarnib in children and young adults with neurofibromatosis type 1 and progressive plexiform neurofibromas. Neuro Oncol. 2014 May;16(5):707-18. doi: 10.1093/neuonc/nou004. Epub 2014 Feb 4. PMID 24500418

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase A -Tipifarnib: Patients receive oral tipifarnib every 12 hours on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.Patients receive tipifarnib ONLY in the first treatment until they progress to the second treatment/crossover to receive placebo.
- Phase B - Placebo: Patients receive oral placebo every 12 hours on days 1-21. Courses repeat as in arm I.Patients receive placebo ONLY in the first treatment until they progress to the second treatment/crossover to receive tipifarnib.
Period: Period 1-First Treatment
Arm/Group | Phase A -Tipifarnib | Phase B - Placebo
Started | 31 | 31 (These are the patients randomized to receive placebo. Two of these patients were deemed ineligible.)
Pts Who Progressed to Second Treatment | 20 | 23
Ineligible Patients | 0 | 2
Completed | 20 | 23
Not Completed | 11 | 8
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Adverse Event | 2 | 1
Not completed — non-adherence | 3 | 0
Not completed — Death | 1 | 0
Not completed — Pts that did not progress | 2 | 2
Not completed — Ineligible | 0 | 2
Period: Period 2-crossover
Arm/Group | Phase A -Tipifarnib | Phase B - Placebo
Started | 20 | 23
Completed | 10 | 12
Not Completed | 10 | 11
Not completed — refused phase B | 2 | 2
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Adverse Event | 2 | 2
Not completed — non-adherence | 1 | 0
Not completed — Pts that did not progress | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Phase A-Tipifarnib: Patients receive oral tipifarnib every 12 hours on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. These are the patients that started on tipifarnib only. This number does not reflect the total amount of patients that crossed over to placebo.
- Phase B - Placebo: Patients receive oral placebo every 12 hours on days 1-21. Courses repeat as in arm I. These are the patients that started on placebo only. This number does not reflect the total amount of patients that crossed over to tipifarnib. Two of the 31 patients were deemed ineligible, thus 29 started placebo.
- Total: Total of all reporting groups
Arm/Group | Phase A-Tipifarnib | Phase B - Placebo | Total
Number analyzed (Participants) | 31 | 31 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 28 | 31 | 59
  Between 18 and 65 years | 3 | 0 | 3
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.2 (5.13) | 9.8 (4.69) | 10. (4.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 15 | 25
  Male | 21 | 16 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 29 | 30 | 59
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 3 | 4 | 7
  White | 25 | 25 | 50
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
  Hispanic | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31 | 31 | 62

OUTCOME MEASURES:

1. Primary Outcome: Median Time to Progression
Description: Median time to progression is defined as a greater than or equal to 20% increase increase in the sum of the volume of all index lesions based on volumetric analysis utilizing magnetic resonance imaging (MRI).Start of phase A or phase B to time of progression.
Time Frame: 8 years
Population: phase A - 62 started and 2 were ineligible = 60 phase B - 43 started
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Phase A - Tipifarnib: Tipifarnib
- Phase B - Placebo: Placebo
Arm/Group | Phase A - Tipifarnib | Phase B - Placebo
Number analyzed (Participants) | 60 | 43
Months
  Placebo | 10.6 [8.1 to 18.3] | 14.5 [8.2 to 26.1]
  Tipifarnib | 19.2 [8.1 to 30.3] | 13.3 [8.0 to 19.6]

2. Primary Outcome: Number of Participants With Adverse Events
Description: Here are the number of participants with adverse events. For the detailed list of adverse events see the adverse event module.
Time Frame: 8 years
Population: Adverse event data is in compliance with DSMB (Data Safety Monitoring Board).
Measure: Count of Participants; unit: Participants
Groups:
- Tipifarnib & Placebo: Patients receive oral tipifarnib every 12 hours on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Patients receive oral placebo every 12 hours on days 1-21. Courses repeat as in arm I.
Arm/Group | Tipifarnib & Placebo
Number analyzed (Participants) | 60
Participants | 59

3. Secondary Outcome: Quality of Life (QOL)
Description: Parents of participants aged 6-18 years completed the Impact of Pediatric Illness (IPI) Scale about their child prior to the start of cycles 1, 4, 7, and 10 and then after every 6 cycles. The IPI Scale assesses QOL in 4 domains: adaptive behavior, emotional functioning, medical/physical status, and cognitive functioning. Responses to the 43 items are made on a 5-point Likert scale (1-5) ranging from "not al all" to "a lot". Higher mean scores indicate better QOL. Parent total scores for participants on placebo were compared with scores from participants receiving tipifarnib on phase A.
Time Frame: Baseline to pre cycle 4
Population: Participants analyzed includes only those whose parents completed the IPI Scale at baseline and pre cycle 4 on phase A.
Measure: Mean (Standard Deviation); unit: Total scores on a scale
Groups:
- Phase A - Tipifarnib: Patients receive oral tipifarnib every 12 hours on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Phase B - Placebo: Patients receive oral placebo every 12 hours on days 1-21. Courses repeat as in arm I.
Arm/Group | Phase A - Tipifarnib | Phase B - Placebo
Number analyzed (Participants) | 18 | 17
Total scores on a scale
  Baseline | 3.69 (0.43) | 3.70 (0.53)
  Pre cycle 4 | 3.91 (0.50) | 3.68 (0.53)
Statistical Analysis 1: Comparison: Phase A - Tipifarnib vs Phase B - Placebo; Test type: Superiority; p = 0.012, Repeated measures ANOVA
Statistical Analysis 2: Comparison: Phase A - Tipifarnib; Post hoc test: tipifarnib group F=7.40; Test type: Other; p = 0.015, Repeated measures ANOVA
Statistical Analysis 3: Comparison: Phase B - Placebo; Post hoc test: placebo group F=0.19; Test type: Other; p = 0.66, Repeated measures ANOVA

4. Other Pre Specified Outcome: Median Time to Progression Using the Conventional 1-Dimensional Response Evaluation Criteria in Solid Tumors (RECIST) Method
Description: Median time to progression is defined as ≥20% increase in diameter based on volumetric analysis using the 1-dimensional RECIST method. Start of phase A or phase B to time of progression.
Time Frame: 8 years
Population: Phase B - Placebo group is not shown because this outcome measure only applies to the Phase A - Tipifarnib group.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase A - Tipifarnib
Number analyzed (Participants) | 1
Months | NA — TTP was not reached because only one patient met criteria for progressive disease (e.g. insufficient number of participants to calculate TTP per protocol).

5. Other Pre Specified Outcome: Median Time to Progression Using the 2-Dimensional World Health Organization (WHO) Solid Tumor Method
Description: Median time to progression is defined as ≥25% increase in area based on volumetric analysis using the 2-dimensional WHO solid tumor method.
Time Frame: 8 years
Population: Phase B- Placebo group is not shown because this outcome measure only applies to the Phase A - Tipifarnib group.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase A - Tipifarnib
Number analyzed (Participants) | 60
Months | 52.5 [36.3 to 52.5]

ADVERSE EVENTS:
Time Frame: 8 years
Description: Adverse event data is in compliance with DSMB(Data Safety Monitoring Board).
Arm/Group | Tipifarnib & Placebo
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 9/60
Other Adverse Events (participants affected / at risk) | 59/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tipifarnib & Placebo (N=60)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Hallucinations (Psychiatric disorders) | 1 (1)
Hypofibrinogenemia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 4 (5)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
SGOT (AST) (Investigations) | 1 (1)
SGPT (ALT) (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tipifarnib & Placebo (N=60)
Abdominal pain (Gastrointestinal disorders) | 20 (26)
Alkaline phosphatase (Metabolism and nutrition disorders) | 2 (2)
Allergic rhinitis (Immune system disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Anorexia (Gastrointestinal disorders) | 10 (11)
Anxiety (Psychiatric disorders) | 1 (1)
Bicarbonate (Metabolism and nutrition disorders) | 17 (21)
Bilirubin (Hepatobiliary disorders) | 8 (9)
Blurred vision (Eye disorders) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Chest pain (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 7 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Creatinine (Investigations) | 3 (3)
Depression (Psychiatric disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 28 (33)
Dizziness (Nervous system disorders) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 2 (2)
Edema (General disorders) | 2 (2)
Flushing (Vascular disorders) | 1 (1)
Hallucinations (Psychiatric disorders) | 1 (1)
Headache (Nervous system disorders) | 11 (16)
Hematuria (Renal and urinary disorders) | 6 (7)
Hemoglobin (Blood and lymphatic system disorders) | 16 (19)
Hemorrhage/bleeding (Blood and lymphatic system disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 5 (5)
Hyperglycemia (Metabolism and nutrition disorders) | 7 (7)
Hyperkalemia (Metabolism and nutrition disorders) | 8 (9)
Hypermagnesemia (Metabolism and nutrition disorders) | 9 (10)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 9 (11)
Hypocalcemia (Metabolism and nutrition disorders) | 7 (8)
Hypofribrinogenemia (Investigations) | 5 (6)
Hypoglycemia (Metabolism and nutrition disorders) | 7 (8)
Hypokalemia (Metabolism and nutrition disorders) | 6 (6)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 9 (9)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (3)
Insomnia (Psychiatric disorders) | 4 (4)
Leukopenia (Investigations) | 1 (1)
Lymphopenia (Investigations) | 12 (14)
Mood alteration-anxiety (Psychiatric disorders) | 3 (3)
Mood alteration-depression (Psychiatric disorders) | 1 (1)
Mouth dryness (Gastrointestinal disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 30 (37)
Neuropathy motor (Nervous system disorders) | 1 (1)
Neuropathy sensory (Nervous system disorders) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 13 (16)
Otalgia (Ear and labyrinth disorders) | 1 (1)
Pain (neck) (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain hands and feet (Musculoskeletal and connective tissue disorders) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2)
Personality/behavioral (Psychiatric disorders) | 1 (1)
Pharyngitis (Infections and infestations) | 2 (2)
Platelets (Investigations) | 8 (9)
Prolonged PT (Investigations) | 26 (33)
Prolonged PTT (Investigations) | 25 (33)
Proteinuria (Renal and urinary disorders) | 12 (12)
Pruritis (Skin and subcutaneous tissue disorders) | 8 (8)
Rash (Skin and subcutaneous tissue disorders) | 14 (16)
Seizure (Nervous system disorders) | 1 (1)
SGOT (AST) (Investigations) | 10 (13)
SGPT (ALT) (Investigations) | 8 (11)
Taste disturbance (Gastrointestinal disorders) | 2 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 24 (28)
white blood cell (WBC) (Investigations) | 23 (26)
Weight loss (Investigations) | 3 (3)
Fatigue (General disorders) | 10 (12)
Fever (Investigations) | 2 (2)
Fibrinogen (Blood and lymphatic system disorders) | 7 (7)
Facial flushing (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2009-06-05): https://cdn.clinicaltrials.gov/large-docs/41/NCT00021541/Prot_SAP_ICF_000.pdf